CLINICAL TRIAL: NCT06299878
Title: Neoadjuvant Monotherapy With Anti-PD1 Agents in Patients With Resectable Stage IIIB-D Melanoma: Analysis of Novel Biomarkers
Brief Title: MelPRO-0322 (CRISTINA Trial) [miCrobiome pRedIctS aPD1 effecTivnes In melaNoma pAtietns]
Acronym: CRISTINA
Status: Recruiting | Type: Observational
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Igor Samoylenko, Senior researcher, MD, PhD, Russian Academy of Medical Sciences
Other Study IDs: MelPRO-0322
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Melanoma, Skin; Melanoma Stage Iii
Keywords: neoadjuvant therapy; stage IIIB-D resectable melanoma; gut microbiota
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — formalin fixed paraffin embedded tissue tumor blocks faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Neoadjuvant
  Interventions: Diagnostic Test: Gut microbiota analysis

INTERVENTIONS:
Diagnostic Test: Gut microbiota analysis — Patients with resectable stage IIIB-D melanoma will have a lymph node core biopsy to confirm metastatic lesions, following standard procedures. Additionally, a portion of the tumor tissue will be preserved for biomarker analysis. Participants will then be instructed to submit fecal samples and complete a dietary questionnaire before receiving three doses of PD1 monotherapy, in accordance with the center's routine practice, typically spanning 6-10 weeks. Between weeks 10 and 12, a radiological assessment of the response will be conducted. Following this, participants will undergo regional lymphadenectomy, and the pathological response will be evaluated. After surgery, patients will be placed on adjuvant therapy for 12 months as per routine practice of the center . Subsequently, they will be monitored for five years, adhering to the institution's standard follow-up protocol.

SUMMARY:
The goal of this observational study is to learn about if new biomarkers such as gut microbiota and molecular genetics melanoma features could predict clinical radiological and pathological response to neoadjuvant monotherapy with anti-PD1 agents in patients with resectable stage IIIB-D melanoma. The main questions it aims to answer are:

* radiological and pathological response rate to three doses of antiPD1 agents;
* do radiological and pathological responses correlate with gut microbiota and melanoma molecular genetics features Participants will receive three doses of aPD1 monotherapy as per center routine practice and will undergo regional lymphadenectomy. Before treatment initiation patients will be asked to bring faeces probes and fill out dietary questionnaire as well as just before the surgery.

After sugery adjuvant therapy will be prescribed for 12 month and patients will be followed up according to institutional routine practice for 5 years.

DETAILED DESCRIPTION:
The clinical efficacy of PD1 inhibitors on the 2-year recurrence-free survival of patients with resectable stage III B-D melanoma will be assessed. This indicator will be compared with a historical control group using adjuvant PD1 immunotherapy and targeted therapy. Various factors will be analyzed for their potential impact on immunotherapy effectiveness, including demographics, disease stage and sub-stage, molecular-genetic status of the tumor, composition of the tumor's lymphoid infiltrate, LDH levels, gut microbiome composition, radiological and pathological response to treatment, and the development of immune-mediated adverse events. These findings may help optimize treatment by implementing neoadjuvant therapy for stage III B-D cutaneous melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Performance status according to the Eastern Cooperative Oncology Group (ECOG) of 0-1.
* Patients who have not previously received immunotherapy with anti-PD1, anti-PDL1, or anti-CTLA4 agents.
* Clinical stage III (B-D), i.e., with clinically or radiologically determined metastatic changes in lymph nodes.
* Histologically confirmed involvement of regional lymph nodes.
* Lesions assessable by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Exclusion Criteria:

* Patients with melanoma of non-skin localizations.
* Patients with active autoimmune diseases.
* Patients with active infectious diseases.
* Patients with severe concomitant diseases with an ECOG status >1.
* Pregnant or lactating patients.
* Patients requiring the intake of glucocorticoids at a dose greater than 10 mg of prednisone (or equivalent) per day.
* Patients requiring the use of, or having received, systemic antibiotics within 4 weeks prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No specific requurements to study population
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival | time from surgery and up to 2 years follow up
  2-year disease-free survival: time from surgery to disease recurrence (either locoregional or distant) or death from any cause

SECONDARY OUTCOMES:
pathological response rate | from enrollment to surgery (in average up to 20 weeks)
  Rate of pathological complete response, near-to-pCR, non-pCR/disease progression

OTHER OUTCOMES:
biomarker reproducibility | from enrollment to end of the study follow up (in average during 6 months since randomization)
  Gut microbiota isolation and 16S-RNA clusterization

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, skin tumor department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
IPD data could be aggregated later with another neoadjuvant study